CLINICAL TRIAL: NCT07394712
Title: Comprehensive Maintenance Program: a Health Haven for COPD in Lleida.The NAPOLEON Project.
Acronym: NAPOLEON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Jessica González Gutiérrez MD, PhD, Clinical Professor, Institut de Recerca Biomèdica de Lleida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIC-3295
Record Dates: First submitted 2025-09-10; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: COPD - Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Randomised Controlled Trial
Keywords: Pulmonary rehabilitation; chronic obstructive pulmonary disease (COPD); Randomised controlled trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding: Role separation will allow for blinding of the outcome assessor and personnel involved in data analysis and interpretation of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised multidimensional pulmonary rehabilitation maintenance program (Experimental): Participants assigned to the intervention group will engage in a supervised, multidimensional pulmonary rehabilitation maintenance program over a period of three months. This program will consist of two weekly sessions of supervised exercise and a total of six educational sessions, each lasting approximately 20 minutes, delivered twice per month. The educational sessions will address key topics such as the prevention and management of chronic obstructive pulmonary disease (COPD) exacerbations and the adoption of healthy lifestyle behaviors. All sessions will be conducted at a comprehensive healthcare center by a physiotherapist who serves as both the program facilitator and case manager. The aim of this intervention is to sustain the clinical benefits achieved during the initial 8-week pulmonary rehabilitation program and to promote long-term self-management and functional capacity.
  Interventions: Behavioral: Interdisciplinary intervention
- Standard physical activity recommendations and unsupervised home exercise (No Intervention): The control group will receive general recommendations for physical activity and a table of exercises to be performed at home, as established in standard clinical practice. They will not receive supervised interventions, however, they will be followed during the 12 months of the study and evaluated at the same times and with the same variables as the intervention group (baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3)).

INTERVENTIONS:
Behavioral: Interdisciplinary intervention — This intervention integrates a structured, interdisciplinary educational and physical activity approach specifically designed for individuals with COPD who have completed a standard pulmonary rehabilitation program. The program is distinguished by its incorporation of six monthly educational sessions addressing key lifestyle-related topics, including sleep hygiene, nutrition based on the Mediterranean diet, smoking cessation, alcohol reduction, and clinical self-management.
  In parallel, participants engage in twice-weekly exercise sessions tailored to their individual capacity, combining aerobic, strength, and functional training. Exercise intensity is prescribed based on initial functional assessments, at 50-80% of the average speed achieved in the six-minute walk test or the workload reached in an incremental cycle ergometer test. All sessions are supervised by physiotherapists and emphasize patient empowerment, behavioral change, and long-term disease management
  Arms: Supervised multidimensional pulmonary rehabilitation maintenance program

SUMMARY:
Introduction:

Pulmonary rehabilitation programs (PRPs) are known to reduce symptoms such as dyspnea and fatigue, while improving functional capacity and quality of life in individuals with chronic obstructive pulmonary disease (COPD). However, the benefits of an initial pulmonary rehabilitation program (PRP) tend to diminish rapidly over time, prompting the development of strategies to maintain these effects. Such strategies include supervised exercise programs, telephone follow-ups, and home-based exercise regimens. Nevertheless, the optimal maintenance strategy remains uncertain.

Objectives:

The primary objective is to evaluate the impact of a supervised, multidimensional maintenance PRP on symptoms and quality of life in individuals with COPD. Additionally, the study aims to compare exercise capacity, healthcare resource utilization, economic benefits, and participant perceptions between the intervention and control groups.

Methodology:

A 12-month randomized controlled trial (RCT) with two parallel groups will be conducted in adults with COPD who have completed an initial 8-week PRP. Participants will be randomly assigned in a 1:1 ratio to either the intervention or control group. The intervention group will undergo a maintenance PRP consisting of two weekly supervised exercise sessions and monthly educational sessions on COPD in a comprehensive health center over a 3-month period. The control group will receive standard clinical care recommendations regarding physical activity. Clinical evaluations will be conducted at four time points throughout the study: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3). Full pulmonary function tests and anthropometric assessments will be performed at T0 and T3. Other variables, including symptom burden, quality of life, functional capacity, mental health, physical activity, sleep-wake pattern, and healthcare utilization, will be systematically collected at all four time points.

DETAILED DESCRIPTION:
Justification Pulmonary rehabilitation programs (PRPs) are a cost-effective therapeutic strategy to reduce dyspnea, improve exercise tolerance, and enhance health-related quality of life in individuals with chronic obstructive pulmonary disease (COPD). Conventional PRPs typically last between 6 and 8 weeks and include physical training, education, and psychosocial support. However, multiple studies have shown that the benefits gained tend to diminish within 3 to 6 months after the initial program ends, especially when structured follow-up and maintenance strategies are not implemented.

In response to this issue, various post-PRP maintenance program modalities have been proposed, such as supervised or unsupervised home-based programs, periodic telephone follow-ups, or group exercise sessions. Despite promising results from some clinical trials, the evidence remains heterogeneous and limited, both in terms of clinical efficacy and feasibility within public health systems. International clinical practice guidelines have emphasized the urgent need to evaluate sustainable and economically viable strategies to maintain the benefits of PRPs, particularly in contexts where structured continuity of care is not guaranteed.

The present study involves the implementation of a supervised maintenance post-pulmonary rehabilitation program (PRP) in an outpatient setting, adequately equipped for the intervention and coordinated by a physiotherapist affiliated with a specialized clinical setting. This intervention will consist of a three-month interdisciplinary maintenance program with biweekly supervised physical exercise sessions, education on COPD and healthy lifestyle habits, and strategies for early detection of exacerbations. It is designed as a randomized controlled trial (RCT) with a 12-month follow-up and clinical evaluations at baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3).

Specific Objectives

1. To compare general and COPD-specific health-related quality of life between intervention and control groups at T0, T1, T2, and T3 using the EuroQol-5 Dimensions questionnaire (EQ-5D) and the COPD Assessment Test (CAT).
2. To assess the impact of the intervention on mental health by comparing anxiety and depression levels between groups at T0, T1, T2, and T3, measured with the Hospital Anxiety and Depression Scale (HADS).
3. To compare functional and exercise capacity between groups at T0, T1, T2, and T3, based on spirometry values, the six-minute walk test (6MWT), and handgrip strength.
4. To compare self-reported physical activity levels using the short version of the International Physical Activity Questionnaire (IPAQ) across time points.
5. To evaluate the sleep-wake pattern and determine the intervention's effect on its modulation, through analysis of sleep-wake pattern and activity variables (total sleep time, sleep latency, wake after sleep onset, light and deep sleep stages) recorded by wearable devices throughout the follow-up.
6. To compare healthcare utilization at T3, including non-hospitalized exacerbations, hospital admissions, and total hospitalization days between groups.
7. To assess the cost-effectiveness of the intervention from the healthcare system perspective, considering direct healthcare-related costs and the clinical benefits achieved.

Study Design This study will be conducted as a 12-month randomized controlled trial (RCT) with four clinical assessment visits, involving two parallel groups of adults diagnosed with chronic obstructive pulmonary disease (COPD) who have completed an initial eight-week PRP. Clinical evaluations will take place at four time points: baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3). Comprehensive pulmonary function tests and anthropometric measurements will be performed at T0 and T3. Other variables (symptoms, quality of life, functional capacity, mental health, physical activity, sleep-wake pattern, and healthcare utilization) will be assessed at all four time points. Participants will be randomly assigned in a 1:1 ratio to either the intervention or control group. The intervention group will attend two weekly supervised exercise sessions and two monthly educational sessions at a public health-affiliated center for three months. The control group will receive general physical activity recommendations in line with standard clinical practice. Clinical assessments will be conducted at T0, T1, T2, and T3, covering respiratory symptoms, health-related quality of life, functional capacity, and healthcare service use.

No booster phase is planned beyond the three-month intervention, as one of the study's secondary objectives is to explore the duration of maintenance PRP effects post-intervention. This will help determine whether clinical, functional, and sleep-wake pattern benefits persist in the medium and long term without continued intervention.

The program includes six educational sessions (20 minutes each), delivered monthly over three months and structured into six key thematic areas:

1. Knowledge about chronic obstructive pulmonary disease (COPD).
2. How dyspnea affects us and how to control it.
3. Importance of physical activity and exercise.
4. Malnutrition and obesity in chronic obstructive pulmonary disease (COPD).
5. Good sleep hygiene is important.
6. Smoking and alcohol cessation.

Adverse Events: Any adverse events observed during the intervention that led to exercise discontinuation will be recorded in an Adverse Event Report Form by the session physiotherapist and reported to the trial's coordinating physiotherapist. As previously stated, if exacerbations are detected, the patient will be referred to the hospital's specialized chronic obstructive pulmonary disease (COPD) clinic. Moreover, as outlined in Table 2, Section 6 (Supervision and Safety), the protocol includes professional supervision during the intervention, individualized adaptation and ongoing monitoring, and supplemental oxygen therapy if necessary.

Randomization: Patients will be randomized 1:1 into two study groups using a sequence generated by an electronic system external to the research team. The randomization sequence will remain concealed from the investigators until an eligible patient has provided written informed consent. Investigators will have secure, password-protected access to the system 24/7.

Blinding: Role separation will allow for blinding of the outcome assessor and personnel involved in data analysis and interpretation of treatment allocation.

Clinical and Functional Variable Evaluation Timeline: Clinical assessments will occur at baseline (T0), 3 months (T1), 6 months (T2), and 12 months (T3). Full spirometry and anthropometric measurements will be conducted at T0 and T3. All other variables (symptoms, quality of life, functional capacity, mental health, physical activity, sleep-wake pattern, and healthcare use) will be assessed at each time point. These include clinical characteristics of chronic obstructive pulmonary disease (COPD) (total number of exacerbations and hospitalizations, and events during the previous year); respiratory symptoms using the Dyspnea-12 questionnaire; mental health via the Hospital Anxiety and Depression Scale (HADS); general quality of life through the EuroQol-5 Dimensions questionnaire (EQ-5D) and COPD-specific quality of life with the COPD Assessment Test (CAT); aerobic capacity via the six-minute walk test (6MWT); handgrip strength using dynamometry; and physical activity levels via the short form of the International Physical Activity Questionnaire (IPAQ). The sleep-wake pattern will be continuously monitored over the 12-month follow-up using wrist-worn devices in both groups to analyze key sleep variables. Adherence to the intervention will be assessed by calculating average session attendance at T3, as will healthcare resource use.

Cost-Effectiveness Analysis: Cost-effectiveness analysis will be conducted using the intention-to-treat principle. Costs during the 12-month study period will be evaluated for both groups. The analysis will adopt a healthcare system perspective, focusing exclusively on patient health outcomes and direct provider-borne costs. The time horizon is 12 months, and all costs will be reported in 2025 euros (€). The intervention's impact on quality of life will be estimated through quality-adjusted life years (QALYs), based on the Health Utilities Index (HUI) derived from EuroQol-5 Dimensions questionnaire (EQ-5D), using the formula: QALYs = 0.5 × baseline HUI + 0.5 × 12-month HUI.

To manage missing data, multiple imputation will be applied independently using the Multivariate Imputation by Chained Equations (MICE) method with predictive mean matching. Initially, the database will be stratified by treatment group to ensure group-specific imputations. The imputation process will include costs, Health Utilities Index (HUI), age, sex, and body mass index (BMI).

To illustrate uncertainty in cost-effectiveness outcomes, 5,000 nonparametric bootstrap replications of cost and effectiveness pairs will be simulated. Pooled cost-effectiveness estimates will be calculated using Rubin's rules and plotted on a cost-effectiveness plane.

Sample Size: Sample size was calculated based on the primary outcome, Dyspnea-12. A clinically relevant difference of 2.83 points at 12-month follow-up was considered. Assuming a common standard deviation of 5 points, a significance level of 0.05, 80% statistical power, and a 10% dropout rate, a total of 43 participants per group is estimated to be required to detect this difference.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 to 75 years.
* Confirmed medical diagnosis of chronic obstructive pulmonary disease (COPD) of moderate to severe severity, based on clinical evaluation and pulmonary function testing.
* Clinically stable for at least 4 weeks following the last severe exacerbation, as confirmed by the treating pulmonologist.
* Referred to an outpatient pulmonary rehabilitation program due to persistent symptoms and a history of exacerbations, with moderate to severe dyspnea (Medical Research Council [MRC] dyspnea scale score > 2), according to physician assessment.
* Completed at least 6 out of 8 sessions of a standard 8-week initial pulmonary rehabilitation program.

Exclusion Criteria:

* Presence of medical contraindications to physical exercise, including unstable cardiovascular conditions (e.g., recent myocardial infarction, uncontrolled arrhythmias), severe musculoskeletal or neurological disorders, recent surgery, or acute medical conditions (e.g., recent stroke) that impair participation.
* Severe cognitive impairment that limits the ability to understand instructions or participate actively in the program.
* Unstable psychiatric disorders that may compromise adherence to or continuity with the exercise regimen.
* Lack of availability or refusal to attend the scheduled sessions of the community-based exercise program.
* Participation in another pulmonary rehabilitation program within the 6 months prior to study enrollment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dyspnea (Dyspnea-12 total score) | Month 12 post-baseline
  Dyspnea will be assessed using the Dyspnea-12 (D-12) questionnaire. The D-12 is a validated self-administered tool that quantifies breathlessness across 12 descriptors (physical and affective). Each item is scored from 0 (none) to 3 (severe), yielding a total score from 0 to 36, with higher scores indicating greater severity. The primary outcome will be the D-12 total score at Month 12, compared between intervention and control groups.

SECONDARY OUTCOMES:
Treatment Adherence (% attendance) | From Baseline to Month 12
  Adherence will be measured as the percentage of attended supervised rehabilitation sessions out of the total prescribed. A threshold of ≥80% will define adequate adherence.
Disease-specific Health-related Quality of Life (COPD Assessment Test, CAT total score) | Baseline, Month 3, Month 6, Month 12
  The CAT is an 8-item validated questionnaire scored 0-40, with higher scores reflecting greater impact of COPD. A change ≥2 points is considered clinically significant.
General Health-related Quality of Life (EQ-5D-5L index and VAS score) | Baseline, Month 3, Month 6, Month 12
  General health-related quality of life will be assessed with the EQ-5D-5L, which includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and a visual analog scale (VAS) from 0 (worst health) to 100 (best health). Utility indices will be calculated to estimate quality-adjusted life years (QALYs) for economic evaluation.
Exercise Capacity (6-minute walk test distance, meters) | Baseline, Month 3, Month 6, Month 12
  Exercise capacity will be measured by total distance walked in the 6-minute walk test, referenced to sex- and age-adjusted norms.
Respiratory Function (FEV1, FVC, DLCO, % predicted) | Baseline, Month 12
  Pulmonary function will be evaluated by spirometry, with results expressed as % predicted based on international reference values.
Direct Healthcare Costs | From Baseline to Month 12
  Direct healthcare costs will be calculated from the healthcare provider perspective, based on hospitalizations, unscheduled visits, and medication use. Costs will be expressed in euros (€) for 2025.
  Unit of Measure: Euros (€)
Quality-adjusted Life Years (QALYs) | From Baseline to Month 12
  QALYs will be estimated using EQ-5D-5L utility scores and area-under-the-curve methods.
  Unit of Measure: QALYs
Cost-utility Ratio | From Baseline to Month 12
  Incremental cost-utility ratios (ICURs) will be calculated by dividing incremental costs (€) by incremental QALYs gained between intervention and control groups. Bootstrapping methods will be used to account for uncertainty.
  Unit of Measure: Incremental cost per QALY (€ / QALY)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Arnau de Vilanova University Hospital, Lleida, Catalonia
  - Arnau de Vilanova University Hospital, Lleida

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying published results, including de-identified data on primary and secondary outcomes, will be made available upon reasonable request. Data will be shared after publication of the main results, for non-commercial academic use, and upon approval of a data-sharing agreement. Supporting documents such as the study protocol and statistical analysis plan will also be available.

REFERENCES:
- [Background] Benjafield A, Tellez D, Barrett M, et al. An estimate of the European prevalence of COPD in 2050. Eur Respir J. 2021;58(suppl 65):OA2866. doi:10.1183/13993003.congress-2021.OA2866
- [Background] Ekstrom MP, Bornefalk H, Skold CM, Janson C, Blomberg A, Bornefalk-Hermansson A, Igelstrom H, Sandberg J, Sundh J. Minimal Clinically Important Differences and Feasibility of Dyspnea-12 and the Multidimensional Dyspnea Profile in Cardiorespiratory Disease. J Pain Symptom Manage. 2020 Nov;60(5):968-975.e1. doi: 10.1016/j.jpainsymman.2020.05.028. Epub 2020 Jun 6. PMID 32512047
- [Background] Gabrio A, Mason AJ, Baio G. Handling Missing Data in Within-Trial Cost-Effectiveness Analysis: A Review with Future Recommendations. Pharmacoecon Open. 2017 Jun;1(2):79-97. doi: 10.1007/s41669-017-0015-6. PMID 29442336
- [Background] Ferro García R, García Ríos MC, Vives Montero MC. Un análisis de la adherencia al tratamiento en fisioterapia. Fisioterapia. 2004;26(6):333-339. doi:10.1016/S0211-5638(04)73120-X
- [Background] Mantilla Toloza SC, Gómez-Conesa A. El Cuestionario Internacional de Actividad Física. Un instrumento adecuado en el seguimiento de la actividad física poblacional. Rev Iberoam Fisioter y Kinesiol. 2007;10(1):48-52. doi:10.1016/S1138-6045(07)73665-1
- [Background] Oteo JA, Benavente P, Garzón M. Valores normativos de la fuerza de puño en la población española en edad laboral. Influencia de las variables antropométricas de la mano y el antebrazo. Rev Iberoam Cirugía la Mano. 2015;43(2):104-110. doi:10.1016/j.ricma.2015.09.005
- [Background] Concha-Cisternas Y, Petermann-Rocha F, Castro-Pinero J, Parra S, Albala C, Wyngard VV, Vasquez J, Cigarroa I, Celis-Morales C. [Handgrip strength as a predictor of adverse health outcomes]. Rev Med Chil. 2022 Aug;150(8):1075-1086. doi: 10.4067/S0034-98872022000801075. Spanish. PMID 37358156
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Agusti A, Fernandez-Villar A, Capelastegui A, Garcia-Losa M, Velasco B, Sanchez G. Validity Study of Catalan, Galician and Basque Language Versions of the COPD Assessment Test and Equivalence With the Spanish Version. Arch Bronconeumol. 2017 Jun;53(6):311-317. doi: 10.1016/j.arbres.2016.10.003. Epub 2016 Dec 13. English, Spanish. PMID 27986409
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Herrero MJ, Blanch J, Peri JM, De Pablo J, Pintor L, Bulbena A. A validation study of the hospital anxiety and depression scale (HADS) in a Spanish population. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):277-83. doi: 10.1016/s0163-8343(03)00043-4. PMID 12850660
- [Background] Amado Diago CA, Puente Maestu L, Abascal Bolado B, Aguero Calvo J, Hernando Hernando M, Puente Bats I, Aguero Balbin R. Translation and Validation of the Multidimensional Dyspnea-12 Questionnaire. Arch Bronconeumol (Engl Ed). 2018 Feb;54(2):74-78. doi: 10.1016/j.arbres.2017.08.001. Epub 2017 Nov 6. English, Spanish. PMID 29122333
- [Background] Agusti A, Celli BR, Criner GJ, Halpin D, Anzueto A, Barnes P, Bourbeau J, Han MK, Martinez FJ, Montes de Oca M, Mortimer K, Papi A, Pavord I, Roche N, Salvi S, Sin DD, Singh D, Stockley R, Lopez Varela MV, Wedzicha JA, Vogelmeier CF. Global Initiative for Chronic Obstructive Lung Disease 2023 Report: GOLD Executive Summary. Am J Respir Crit Care Med. 2023 Apr 1;207(7):819-837. doi: 10.1164/rccm.202301-0106PP. No abstract available. PMID 36856433
- [Background] Gloeckl R, Marinov B, Pitta F. Practical recommendations for exercise training in patients with COPD. Eur Respir Rev. 2013 Jun 1;22(128):178-86. doi: 10.1183/09059180.00000513. PMID 23728873
- [Background] Carneiro-Barrera A, Amaro-Gahete FJ, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Tinahones FJ, Ruiz JR. Effect of a Weight Loss and Lifestyle Intervention on Dietary Behavior in Men with Obstructive Sleep Apnea: The INTERAPNEA Trial. Nutrients. 2022 Jun 30;14(13):2731. doi: 10.3390/nu14132731. PMID 35807913
- [Background] Carneiro-Barrera A, Amaro-Gahete FJ, Saez-Roca G, Martin-Carrasco C, Palmeira AL, Ruiz JR. Interdisciplinary Weight Loss and Lifestyle Intervention for Daily Functioning and Psychiatric Symptoms in Obstructive Sleep Apnea: The INTERAPNEA Randomized Clinical Trial. J Clin Psychiatry. 2023 Jun 12;84(4):22m14502. doi: 10.4088/JCP.22m14502. PMID 37339363
- [Background] Carneiro-Barrera A, Amaro-Gahete FJ, Guillen-Riquelme A, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Buela-Casal G, Ruiz JR. Effect of an Interdisciplinary Weight Loss and Lifestyle Intervention on Obstructive Sleep Apnea Severity: The INTERAPNEA Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e228212. doi: 10.1001/jamanetworkopen.2022.8212. PMID 35452108
- [Background] Ambrosino N, Bertella E. Lifestyle interventions in prevention and comprehensive management of COPD. Breathe (Sheff). 2018 Sep;14(3):186-194. doi: 10.1183/20734735.018618. PMID 30186516
- [Background] Holland AE, Cox NS, Houchen-Wolloff L, Rochester CL, Garvey C, ZuWallack R, Nici L, Limberg T, Lareau SC, Yawn BP, Galwicki M, Troosters T, Steiner M, Casaburi R, Clini E, Goldstein RS, Singh SJ. Defining Modern Pulmonary Rehabilitation. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2021 May;18(5):e12-e29. doi: 10.1513/AnnalsATS.202102-146ST. PMID 33929307
- [Background] Blackstock FC, Lareau SC, Nici L, ZuWallack R, Bourbeau J, Buckley M, Durning SJ, Effing TW, Egbert E, Goldstein RS, Kelly W, Lee A, Meek PM, Singh S; American Thoracic Society, Thoracic Society of Australia and New Zealand, Canadian Thoracic Society, and British Thoracic Society. Chronic Obstructive Pulmonary Disease Education in Pulmonary Rehabilitation. An Official American Thoracic Society/Thoracic Society of Australia and New Zealand/Canadian Thoracic Society/British Thoracic Society Workshop Report. Ann Am Thorac Soc. 2018 Jul;15(7):769-784. doi: 10.1513/AnnalsATS.201804-253WS. PMID 29957038
- [Background] Burns DK, Wilson EC, Browne P, Olive S, Clark A, Galey P, Dix E, Woodhouse H, Robinson S, Wilson A. The Cost Effectiveness of Maintenance Schedules Following Pulmonary Rehabilitation in Patients with Chronic Obstructive Pulmonary Disease: An Economic Evaluation Alongside a Randomised Controlled Trial. Appl Health Econ Health Policy. 2016 Feb;14(1):105-15. doi: 10.1007/s40258-015-0199-9. PMID 26346590
- [Background] Cecins N, Geelhoed E, Jenkins SC. Reduction in hospitalisation following pulmonary rehabilitation in patients with COPD. Aust Health Rev. 2008 Aug;32(3):415-22. doi: 10.1071/ah080415. PMID 18666869
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Spencer LM, McKeough ZJ. Maintaining the benefits following pulmonary rehabilitation: Achievable or not? Respirology. 2019 Sep;24(9):909-915. doi: 10.1111/resp.13518. Epub 2019 Mar 19. PMID 30891887
- [Background] Guell MR, Cejudo P, Ortega F, Puy MC, Rodriguez-Trigo G, Pijoan JI, Martinez-Indart L, Gorostiza A, Bdeir K, Celli B, Galdiz JB. Benefits of Long-Term Pulmonary Rehabilitation Maintenance Program in Patients with Severe Chronic Obstructive Pulmonary Disease. Three-Year Follow-up. Am J Respir Crit Care Med. 2017 Mar 1;195(5):622-629. doi: 10.1164/rccm.201603-0602OC. PMID 27611807
- [Background] Jenkins AR, Gowler H, Curtis F, Holden NS, Bridle C, Jones AW. Efficacy of supervised maintenance exercise following pulmonary rehabilitation on health care use: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2018 Jan 10;13:257-273. doi: 10.2147/COPD.S150650. eCollection 2018. PMID 29391784
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Beauchamp MK, Evans R, Janaudis-Ferreira T, Goldstein RS, Brooks D. Systematic review of supervised exercise programs after pulmonary rehabilitation in individuals with COPD. Chest. 2013 Oct;144(4):1124-1133. doi: 10.1378/chest.12-2421. PMID 23429931
- [Background] Alison JA, McKeough ZJ, Johnston K, McNamara RJ, Spencer LM, Jenkins SC, Hill CJ, McDonald VM, Frith P, Cafarella P, Brooke M, Cameron-Tucker HL, Candy S, Cecins N, Chan AS, Dale MT, Dowman LM, Granger C, Halloran S, Jung P, Lee AL, Leung R, Matulick T, Osadnik C, Roberts M, Walsh J, Wootton S, Holland AE; Lung Foundation Australia and the Thoracic Society of Australia and New Zealand. Australian and New Zealand Pulmonary Rehabilitation Guidelines. Respirology. 2017 May;22(4):800-819. doi: 10.1111/resp.13025. Epub 2017 Mar 24. PMID 28339144
- [Background] Jenkins S, Hill K, Cecins NM. State of the art: how to set up a pulmonary rehabilitation program. Respirology. 2010 Nov;15(8):1157-73. doi: 10.1111/j.1440-1843.2010.01849.x. PMID 20920127
- [Background] Blanco I, Diego I, Bueno P, Casas-Maldonado F, Miravitlles M. Geographic distribution of COPD prevalence in the world displayed by Geographic Information System maps. Eur Respir J. 2019 Jul 18;54(1):1900610. doi: 10.1183/13993003.00610-2019. Print 2019 Jul. No abstract available. PMID 31000678